CLINICAL TRIAL: NCT06987097
Title: Ambrisentan for the Treatment of Early-Stage Low-Risk Pulmonary Arterial Hypertension: A Multicenter, Randomized, Double-Blind, Placebo-Controlled ALEPH Trial
Brief Title: Ambrisentan for Early Low-Risk Pulmonary Arterial Hypertension
Acronym: ALEPH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hang Zhang, Professor, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY20250327-11
Record Dates: First submitted 2025-04-24; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Arterial Hypertension (PAH)
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ambrisentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambrisentan (Experimental): Monotherapy using ambrisentan will start at a dose of 5 mg (once daily) and will be up-titrated to 10mg (once daily) after 2 weeks apart if patients are tolerable.
  Interventions: Drug: Ambrisentan
- Placebo Placebo tablet (Placebo Comparator): Placebo tablet (one to two tablets corresponding to one to two verum tablets).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ambrisentan — After two weeks of initial treatment, the study drugs' dose will be increased to two tablets per day (10 mg/day). If the patient cannot tolerate the increased dose (e.g., experiencing headache, dizziness, palpitations, hypotension, or other drug-related symptoms or signs), the dose will be reduced to 5 mg/day. If the study drug has reached the maximum allowable dose (two tablets/day) and the patient shows signs of worsening PAH or right heart failure, the clinician may decide to add diuretics (with the type and dosage left at the referring physician's discretion). The number and percentage of patients requiring diuretic combination therapy in both groups will be recorded. Other baseline treatment medications will remain unchanged through follow-up duration.
  Arms: Ambrisentan
Drug: Placebo — Placebo tablet (one to two tablets corresponding to one to two verum tablets). Administration: Placebo will be administrated orally with or without food intake in the morning.
  Arms: Placebo Placebo tablet

SUMMARY:
This is an investigator-initiated, multicenter, randomized, double-blind, placebo-controlled clinical trial.

DETAILED DESCRIPTION:
Early-stage low-risk PAH is defined as mean pulmonary arterial pressure (mPAP) between 20 and 25 mmHg at rest, measured by right heart catheterization, and classified as low-risk based on the 2022 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension. Patients will be randomized at a 1:1 ratio to either the treatment group (Ambrisentan group) or the control group (Placebo group). Treatment group: Ambrisentan, with an initial dose of 5 mg/day (one tablet per day).Control group: Placebo, which will be provided in the same appearance and taste as Ambrisentan, one tablet per day.

After two weeks of initial treatment, the study drugs' dose will be increased to two tablets per day (10 mg/day). If the patient cannot tolerate the increased dose (e.g., experiencing headache, dizziness, palpitations, hypotension, or other drug-related symptoms or signs), the dose will be reduced to 5 mg/day. If the study drug has reached the maximum allowable dose (two tablets/day) and the patient shows signs of worsening PAH or right heart failure, the clinician may decide to add diuretics (with the type and dosage left at the referring physician's discretion). The number and percentage of patients requiring diuretic combination therapy in both groups will be recorded. Other baseline treatment medications will remain unchanged through follow-up duration.

The study drugs will be administered continuously for 12 months, then unblinding will be performed. Thereafter, patients who have reached the primary endpoint must undertake Ambrisentan. For patients who have not reached the primary endpoint, the subsequent medications treatment will be left at the PAH specialist's discretion. Follow-up will be undertaken at the following timing: Month 1, Month 6, and Month 12, with additional follow-up extending up to 3 years. All clinical drugs involved in this study have completed registration for market approval in China and are currently in clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* mPAP > 20 mmHg and < 25 mmHg, pulmonary vascular resistance (PVR) > 2 WUs and ≤ 3 WUs, and pulmonary arterial wedge pressure (PAWP) ≤ 15 mmHg via right heart catheterization (RHC); RHC measurement will be accepted if it was done within 7 days before enrollment;
* Group I PAH, including idiopathic PAH (IPAH), heritable PAH (HPAH), Drug- and toxin-induced PAH, associated with connective tissue disease (connective tissue disease at good control), associated with portal hypertension, associated with congenital heart disease;
* At low risk based on the 2022 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension three-strata risk-assessment model;
* The subject or a legally authorized representative must understand the study requirements, agree to the treatment procedures, and provide written informed consent before any study-specific procedures are performed;
* The subject must demonstrate a willingness and ability to comply with all protocol requirements.

Exclusion Criteria:

* Patients currently receiving PAH specific medications, regardless of whether mPAP is between 20-25 mmHg. PAH specific medications include endothelin receptor antagonists (ERAs; e.g., bosentan, ambrisentan, macitentan), phosphodiesterase type 5 inhibitors (PDE5i; e.g., sildenafil, tadalafil, vardenafil), prostacyclin analogs (e.g., iloprost, epoprostenol, treprostinil, beraprost), soluble guanylate cyclase stimulators (e.g., riociguat). Intermittent use of PDE5 inhibitors for the treatment of male erectile dysfunction is permitted;
* Intolerance to ambrisentan or its excipients;
* Pulmonary veno-occlusive disease (PVOD);
* Pulmonary capillary hemangiomatosis (PCH);
* Within 6 months after congenital heart disease surgical repair or percutaneous closure procedure;
* Group II-V PH;
* Clinically significant anemia, defined as hemoglobin concentration below 75% of the lower limit of normal;
* Renal insufficiency, defined as estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m² within 3 months prior to enrollment;
* Elevated Alanine Aminotransferase （ALT） and/or Aspartate Aminotransferase （AST） exceeding 3 times the upper limit of normal (ULN);
* Systolic blood pressure < 85 mmHg;
* Uncontrolled hypertension, defined as blood pressure > 160/90 mmHg at rest and/or > 220/120 mmHg under stress conditions;
* Participation in any clinical drug trial within 4 weeks prior to screening and/or planned participation in another clinical drug trial during this study;
* Expected life expectancy of less than 1 year;
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the composite of pulmonary hypertension progression at 12 months | baseline,12 months
  defined as meeting any of the following criteria within 12 months:
  1. mPAP ≥ 25 mmHg OR PVR > 3 WUs as measured by RHC OR
  2. worsening of risk stratification compared to baseline, defining as at least one class progression based on the simplified four-tier model of the 2022 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension

SECONDARY OUTCOMES:
systolic PAP (sPAP) by Hemodynamic measurements | baseline,12 months
mPAP by Hemodynamic measurements | baseline,12 months
cardiac output (CO) by Hemodynamic measurements | baseline,12 months
cardiac index (CI) by Hemodynamic measurements | baseline,12 months
PVR by Hemodynamic measurements | baseline,12 months
PVRi by Hemodynamic measurements | baseline,12 months
PAWP by Hemodynamic measurements | baseline,12 months
right atrial pressure by Hemodynamic measurements | baseline,12 months
pulmonary arterial compliance by Hemodynamic measurements | baseline,12 months
diameter of chambers by Echocardiographic measurements | baseline,12 months
ejection fraction by Echocardiographic measurements | baseline,12 months
right ventricular (RV) fraction of area change (FAC) by Echocardiographic measurements | baseline,12 months
TAPSE by Echocardiographic measurements | baseline,12 months
pulmonary artery accelation time (PAAT) by Echocardiographic measurements | baseline,12 months
regurgitation of tricuspid or pulmonary valve by Echocardiographic measurements | baseline,12 months
sPAP by Echocardiographic measurements | baseline,12 months
RAP by Echocardiographic measurements | baseline,12 months
WHO functional class through follow - up | baseline,12 months
Borg index through follow - up | baseline,12 months
N-terminal-pro BNP | baseline,12 months
6-minute walk distance (6MWD) | baseline,12 months
Time to the first occurrence of the following events, analyzed using log-rank and LWYY model | baseline,12 months
  * All-cause mortality
  * Hospitalization due to PAH worsening
  * Clinical deterioration of PAH, defined as the need for diuretics or digoxin (oral or intravenous), or the need of combination therapy with PAH specific medications
  * 6MWD decreases by 10% or 30m

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Liang Chen MD, PhD, Study Chair — Nanjing First Hospital, Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kan JY, Zhang XJ, Yu WD, Yang ZW, Fan FL, Ding GW, Luo J, Li W, Xie DJ, Liu XF, Zhang H, Chen SL. Ambrisentan for Early-Stage Low-Risk Pulmonary Arterial Hypertension: Design of the Randomized, Double-Blind, Placebo-Controlled ALEPH Trial. JACC Asia. 2026 Jan 28:S2772-3747(26)00027-X. doi: 10.1016/j.jacasi.2025.12.014. Online ahead of print. PMID 41653169